CLINICAL TRIAL: NCT02674399
Title: A Phase 2, Double-Blind, Randomized, Controlled Study to Evaluate the Efficacy and Safety of JointStem, Autologous Adipose Tissue Derived Mesenchymal Stem Cells, in Treatment of Osteoarthritis
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of JointStem in Treatment of Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nature Cell Co. Ltd. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-OAP2-US01
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — hylan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JointStem (Experimental): autologous adipose tissue derived mesenchymal stem cells (AdMSC)
  Interventions: Drug: JointStem
- Synvisc-One (Active Comparator): hyaluronic acid
  Interventions: Drug: Synvisc-One

INTERVENTIONS:
Drug: JointStem
  Arms: JointStem
Drug: Synvisc-One
  Other Names: Active Comparator
  Arms: Synvisc-One

SUMMARY:
This study is a double-blind, randomized, controlled study with two arms to evaluate JointStem as a treatment for subjects with osteoarthritis. Following a 2-week screening period, approximately 30 subjects will be randomly assigned into one of the following two arms in a 2:1 ratio (2 JointStem : 1 positive control). After each subject completes 6-month visit (Visit 6) and the data management team confirms all data have no issue, the individual database will be locked and the blinding will be open for the statistical analysis.Only subjects who are assigned will be requested to visit the study center for 9-month and 12-month follow-up visits (Visits 7 and 8). To see long-term effects of JointStem, all subjects who complete Visit 6 will be requested to visit the study center at 24-month after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Subject who can give written informed consent
* Male or female of any race, aged 22-60
* Subject who had osteoarthritis of knee diagnosed at least six months prior to Screening
* Subject who has joint pain ≥ 40mm on VAS (Visual Analog Scale) at Screening
* Subject who has swelling, tenderness and active range of motion ≥ Grade I at Screening
* Subject who seeks invasive interventions of intra-articular injections
* Subject who is willing to discontinue all pain medications for osteoarthritis except rescue medication (< acetaminophen 3.25 g per day) at least 72 hours prior to screening and throughout the duration of study
* Subject who has radiographic evidence of grade 3 to 4 osteoarthritis based on the Kellgren and Lawrence radiographic criteria.
* Female subject who is neither pregnant nor lactating
* Subject who is able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Subject who has Body Mass Index (BMI) > 35 kg/m2
* Subject who has unstable knees
* Subject who took any NSAID within two weeks from Screening
* Subject who had any intra-articular injection therapy in any joint within 2 months from Screening
* Subject who has any clinically significant disease, which is judged by the investigator to affect this clinical trial
* Subject who has inflammatory arthropathy (rheumatoid, psoriatic, or avascular necrosis), and post traumatic or septic arthritis
* Subject who has chondrocalcinosis, Paget's disease, Villonodular synovitis, and other non-OA joint diseases
* Subject who has HIV/viral hepatitis
* Subject who had knee surgery or radiation therapy in the affected joint within 6 months from Screening
* Subject who had CVA attack within 6 months from Screening
* Subject for whom the investigator judges the liposuction can cause any problem
* Subject who has significant lab abnormalities
* Subject who has history of local anesthetic allergy
* Subject who took immunosuppressants such as Cyclosporin A or azathioprine within 6 weeks from Screening
* (If a subject uses aspirin or plavix) Subject for whom it is determined that it would not be safe to stop the aspirin/plavix therapy for 2 weeks prior to Visit 2
* Subject who uses anticoagulants which cannot be stopped or corrected
* Subject who had oral or intra-muscular corticosteroids within 30 days from Visit 2
* Subject who had intra-articular corticosteroid injection in any joint within 30 days from Visit 2
* Subject who had intra-articular hyaluronic acid injection within 30 days from Visit 2
* Subject who has known hypersensitivity (allergy) to hyaluronan (sodium hyaluronate) preparations or gram positive proteins
* Subject who has knee joint infections or skin diseases or infections in the area of the injection site
* Subject who has known systemic bleeding disorders
* Subject who is an active drug/EtOH abuser
* Subject who was enrolled in any other clinical trials within 2 months from Screening
* Subject who the principal investigator considers inappropriate for the study due to any other reasons than those listed above
* Subject whose MRI scan results at screening do not demonstrate any sign of cartilage damage

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orthopedic Pain Specialists, Santa Monica, California
  - Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- JointStem: JointStem : autologous adipose tissue derived mesenchymal stem cells (AdMSC) 1x10e8 cells At Visit 3 (Week 0, baseline), the randomized subject received a single intra-articular injection.
- Synvisc-One: hyaluronic acid At Visit 3 (Week 0, baseline), the randomized subject received a single intra-articular injection.
Period: Overall Study
Arm/Group | JointStem | Synvisc-One
Started | 19 | 9
Completed | 17 | 9
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- JointStem: autologous adipose tissue derived mesenchymal stem cells (AdMSC)
  JointStem
- Synvisc-One: hyaluronic acid
  Synvisc-One
- Total: Total of all reporting groups
Arm/Group | JointStem | Synvisc-One | Total
Number analyzed (Participants) | 19 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (6.98) | 52.1 (9.56) | 52.3 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: cm] | 173.66 (9.222) | 169.46 (10.073) | 172.31 (9.527)
Weight [Mean (Standard Deviation); unit: kg] | 81.31 (14.642) | 71.66 (20.569) | 78.2 (17.01)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.903 (4.1938) | 24.572 (4.6408) | 26.154 (4.3971)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score in JointStem Group
Description: Comparing the baseline and 6-month WOMAC scores in JointStem group Score range: 0-2,400 A score of 2,400 represents the most severe impairment and 0 represents the least impairment
Time Frame: Baseline and 6 months
Population: The primary endpoints were evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale | -20.121 (21.0415) |

2. Primary Outcome: Change From Baseline on Visual Analog Scale (VAS) in JointStem Group
Description: Comparing the baseline and 6-month VAS scores in JointStem group Score range: 0-100 A score of 100 represents the most severe pain and 0 represents the least pain.
Time Frame: Baseline and 6 months
Population: The primary endpoints were evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale | -32.5 (23.93) |

3. Primary Outcome: MRI Improvement Evaluation in JointStem Group
Description: Comparing the baseline and 6-month MRI improvement values in JointStem group MRI Improvement Evaluation was conducted by an MRI analysis company called 'Qmetrics'. The main radiological features evaluated were bone marrow edema, osteophytes, and cartilage. Certain features, such as the appearance of a new cartilage defect or increase in the size of existing cartilage defects or osteophytes, is generally considered an indication of osteoarthritic progression. Similarly, the diminishing in severity or size of existing abnormalities would generally be considered to be a healing(improving) response.
Time Frame: 6 months
Population: The primary endpoints were evaluated only in the JointsStem group. And one patient was excluded from the table due to absence of MRI values.
Measure: Count of Participants; unit: Participants
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 18 | 0
Participants
  Improvement | 5 | 0
  No Change | 5 | 0
  Progress | 8 | 0

4. Secondary Outcome: Change From Baseline on WOMAC Between JointStem and Positive Control Groups
Description: Comparing the changes of WOMAC scores between JointStem and positive control groups at 6 months Score range: 0-2,400 A score of 2,400 represents the most severe impairment and 0 represents the least impairment
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale | -20.505 (3.665) | -17.129 (5.3281)

5. Secondary Outcome: Change From Baseline on VAS Between JointStem and Positive Control Groups
Description: Comparing the changes of VAS scores between JointStem and positive control groups at 6 months Score range: 0-100 A score of 100 represents the most severe pain and 0 represents the least pain.
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale | -31.9 (4.90) | -30.6 (7.13)

6. Secondary Outcome: Change From Baseline on Knee Injury & Osteoarthritis Outcome Score (KOOS) Between JointStem and Positive Control Groups
Description: Comparing the changes of KOOS values between JointStem and positive control groups at 6 months KOOS score = 100 - [{(average score of each item) * 100} / 4 ] Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale
  Symptoms | 9.70 (2.888) | 14.83 (4.22)
  Pain | 21.40 (3.975) | 19.04 (5.78)
  ADL | 18.53 (3.937) | 15.94 (5.72)
  Sport/Rec | 25.00 (5.123) | 26.68 (7.482)
  QOL | 22.68 (5.383) | 11.15 (7.884)

7. Secondary Outcome: Change From Baseline on Lysholm Knee Scoring Scale Between JointStem and Positive Control Groups
Description: Comparing the changes of Lysholm Knee Scoring Scales between JointStem and positive control groups at 6 months Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale | 18.9 (3.97) | 19.9 (5.78)

8. Secondary Outcome: Change From Baseline on International Knee Documentation Committee (IKDC) Between JointStem and Positive Control Groups
Description: Comparing the changes of IKDC scores between JointStem and positive control groups at 6 months IKDC score = {(sum of each item score) / 87} * 100 Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale | 55.74 (2.223) | 54.24 (3.238)

9. Secondary Outcome: Change From Baseline on RAND-36 Score Between JointStem and Positive Control Groups
Description: Comparing the changes of RAND-36 scores between JointStem and positive control groups at 6 months Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 9
score on a scale
  Physical Functioning | 17.2 (3.80) | 14.9 (5.52)
  Role Limitation (Physical) | 20.7 (8.04) | 17.4 (11.73)
  Role Limitation (Emotional) | 6.7 (6.615) | -6.74 (9.654)
  Energy/Fatigue | 5.2 (3.91) | 4.5 (5.76)
  Emotional well-being | -3.4 (2.31) | 0.5 (3.45)
  Social Functioning | 14.71 (2.964) | 16.16 (4.312)
  Pain | 21.59 (4.211) | 14.7 (6.18)
  General Health | 2.91 (2.516) | 3.13 (3.668)

10. Secondary Outcome: Change From Baseline on WOMAC in JointStem Group
Description: Comparing the baseline and 9-month/12-month WOMAC scores in JointStem group Score range: 0-2,400 A score of 2,400 represents the most severe impairment and 0 represents the least impairment
Time Frame: Baseline, 9 months and 12 months
Population: This measure was evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 9 | -21.216 (20.9653) |
  Change from baseline at Month 12 | -21.711 (19.7521) |

11. Secondary Outcome: Change From Baseline on VAS in JointStem Group
Description: Comparing the baseline and 9-month/12-month VAS scores in JointStem group Score range: 0-100 A score of 100 represents the most severe pain and 0 represents the least pain.
Time Frame: Baseline, 9 months and 12 months
Population: This measure was evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 9 | -31.5 (25.52) |
  Change from baseline at Month 12 | -35 (24.56) |

12. Secondary Outcome: Comparison of MRI Improvement Evaluation in JointStem Group
Description: Comparing the baseline and 9-month/12-month MRI improvement values in JointStem group MRI Improvement Evaluation was conducted by an MRI analysis company called 'Qmetrics'. The main radiological features evaluated were bone marrow edema, osteophytes, and cartilage. Certain features, such as the appearance of a new cartilage defect or increase in the size of existing cartilage defects or osteophytes, is generally considered an indication of osteoarthritic progression. Similarly, the diminishing in severity or size of existing abnormalities would generally be considered to be a healing(improving) response.
Time Frame: Baseline, 6 months and 12 months
Population: This measure was evaluated only in the JointsStem group. And one patient was excluded from the table due to absence of MRI values.
Measure: Count of Participants; unit: Participants
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 18 | 0
Participants
  Month 6 Improved -> Month 12 Improved | 3 |
  Month 6 Improved -> Month 12 No Change | 1 |
  Month 6 Improved -> Month 12 Progress | 1 |
  Month 6 No Change -> Month 12 Improved | 1 |
  Month 6 No Change -> Month 12 No Change | 2 |
  Month 6 No Change -> Month 12 Progress | 2 |
  Month 6 Progress -> Month 12 Improved | 2 |
  Month 6 Progress -> Month 12 No Change | 0 |
  Month 6 Progress -> Month 12 Progress | 6 |

13. Secondary Outcome: Change of Lysholm Knee Scoring Scale From Baseline at Months 6, 9 and 12
Description: Comparing the baseline and 6-month/9-month/12-month Lysholm Knee Scoring Scale in JointStem group Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: Baseline, 6 months, 9 months and 12 months
Population: This measure was evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 6 | 18.3 (22.29) |
  Change from baseline at Month 9 | 16.1 (25.34) |
  Change from baseline at Month 12 | 17.1 (23.78) |

14. Secondary Outcome: Change of KOOS Score From Baseline at Month 6, 9 and 12 for JointStem Group
Description: Comparing the baseline and 6-month/9-month/12-month KOOS scores in JointStem group KOOS score = 100 - [{(average score of each item) * 100} / 4 ] Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: baseline, 6 month, 9 month, 12 month
Population: This measure was evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 6 (Symptoms) | 9.02 (15.381) |
  Change from baseline at Month 9 (Symptoms) | 15.03 (13.677) |
  Change from baseline at Month 12 (Symptoms) | 15.41 (18.229) |
  Change from baseline at Month 6 (Pain) | 21.65 (20.386) |
  Change from baseline at Month 9 (Pain) | 23.98 (23.200) |
  Change from baseline at Month 12 (Pain) | 25.31 (21.219) |
  Change from baseline at Month 6 (ADL) | 18.66 (23.842) |
  Change from baseline at Month 9 (ADL) | 18.42 (25.017) |
  Change from baseline at Month 12 (ADL) | 21.90 (23.237) |
  Change from baseline at Month 6 (Sport/Rec) | 25.53 (23.915) |
  Change from baseline at Month 9 (Sport/Rec) | 28.42 (25.279) |
  Change from baseline at Month 12 (Sport/Rec) | 33.68 (24.486) |
  Change from baseline at Month 6 (QOL) | 23.36 (24.829) |
  Change from baseline at Month 9 (QOL) | 29.95 (27.228) |
  Change from baseline at Month 12 (QOL) | 28.96 (29.121) |

15. Secondary Outcome: Change of IKDC Score From Baseline at Month 6, 9 and 12 for JointStem Group
Description: Comparing the baseline and 6-month/9-month/12-month IKDC scores in JointStem group IKDC score = {(sum of each item score) / 87} * 100 Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: baseline, 6 month, 9 month, 12 month
Population: This measure was evaluated only in the JointsStem group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 6 | 7.03 (11.379) |
  Change from baseline at Month 9 | 10.95 (12.047) |
  Change from baseline at Month 12 | 9.63 (10.380) |

16. Secondary Outcome: Change of RAND-36 Score From Baseline at Month 6, 9 and 12 for JointStem Group
Description: Comparing the baseline and 6-month/9-month/12-month RAND-36 scores in JointStem group Score range: 0-100 A score of 0 represents the most severe impairment and 100 represents the least impairment
Time Frame: baseline, 6 month, 9 month, 12 month
Population: This measure was evaluated only in the JointsStem group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JointStem | Synvisc-One
Number analyzed (Participants) | 19 | 0
score on a scale
  Change from baseline at Month 6 (Physical Functioning) | 17.4 (22.13) |
  Change from baseline at Month 9 (Physical Functioning) | 18.7 (23.38) |
  Change from baseline at Month 12 (Physical Functioning) | 17.1 (28.69) |
  Change from baseline at Month 6 (Role Limitation_Physical) | 22.4 (36.22) |
  Change from baseline at Month 9 (Role Limitation_Physical) | 30.3 (38.71) |
  Change from baseline at Month 12 (Role Limitation_Physical) | 31.6 (40.69) |
  Change from baseline at Month 6 (Role Limitation_Emotional) | 8.77 (33.048) |
  Change from baseline at Month 9 (Role Limitation_Emotional) | 7.02 (30.604) |
  Change from baseline at Month 12 (Role Limitation_Emotional) | 8.77 (33.048) |
  Change from baseline at Month 6 (Energy/Fatigue) | 2.9 (20.70) |
  Change from baseline at Month 9 (Energy/Fatigue) | 5.3 (16.45) |
  Change from baseline at Month 12 (Energy/Fatigue) | 7.6 (18.81) |
  Change from baseline at Month 6 (Emotional well-being) | -3.4 (10.61) |
  Change from baseline at Month 9 (Emotional well-being) | -3.6 (11.31) |
  Change from baseline at Month 12 (Emotional well-being) | -4.0 (14.79) |
  Change from baseline at Month 6 (Social Functioning) | 13.82 (23.531) |
  Change from baseline at Month 9 (Social Functioning) | 14.47 (20.943) |
  Change from baseline at Month 12 (Social Functioning) | 7.24 (25.109) |
  Change from baseline at Month 6 (Pain) | 23.16 (21.982) |
  Change from baseline at Month 9 (Pain) | 23.95 (22.100) |
  Change from baseline at Month 12 (Pain) | 24.34 (21.967) |
  Change from baseline at Month 6 (General Health) | 3.51 (13.566) |
  Change from baseline at Month 9 (General Health) | 5.71 (10.502) |
  Change from baseline at Month 12 (General Health) | 2.85 (18.636) |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | JointStem | Synvisc-One
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/9
Other Adverse Events (participants affected / at risk) | 18/19 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JointStem (N=19) | Synvisc-One (N=9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 0
Stiff knees (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Injection site pain (General disorders) | 9 | 1
Injection site swelling (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT02674399/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT02674399/SAP_001.pdf
  • Informed Consent Form (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT02674399/ICF_002.pdf